CLINICAL TRIAL: NCT03272425
Title: A Randomized, Open-label, Replicate, Crossover, 4-period Study to Assess the Bioequivalence of Lesinurad/Allopurinol Fixed-dose Combination 200/300 mg Tablets From Ardea Biosciences, Inc. (Test Drug) Versus Lesinurad, 200 mg Tablet From AstraZeneca (Comparator 1) Coadministered With Zyloric®, Allopurinol 300 mg Tablet From Aspen Pharma Industria Farmaceutica Ltda. (Comparator 2) in Healthy Female and Male Adult Subjects, Under Fasting Conditions.
Brief Title: Lesinurad/Allopurinol 200/300 Fixed-Dose Combination (FDC) Tablets Bioequivalence.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ardea Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RDEA594-504
Record Dates: First submitted 2017-09-01; First posted 2017-09-05 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Gout
MeSH Terms: conditions — Gout | interventions — lesinurad; Allopurinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sequence ABBA (Experimental): Treatment A: Lesinurad/Allopurinol FDC Tablets - 200/300 mg (test product); Treatment B: lesinurad, tablets, 200 mg + Zyloric®, allopurinol, tablet, 300 mg (comparator 1 + comparator 2).
  Interventions: Drug: lesinurad/allopurinol 200/300 FDC tablets; Drug: lesinurad 200 mg; Drug: allopurinol 300 mg
- Sequence BABA (Experimental): Treatment A: Lesinurad/Allopurinol FDC Tablets - 200/300 mg (test product); Treatment B: lesinurad, tablets, 200 mg + Zyloric®, allopurinol, tablet, 300 mg (comparator 1 + comparator 2).
  Interventions: Drug: lesinurad/allopurinol 200/300 FDC tablets; Drug: lesinurad 200 mg; Drug: allopurinol 300 mg
- Sequence ABAB (Experimental): Treatment A: Lesinurad/Allopurinol FDC Tablets - 200/300 mg (test product); Treatment B: lesinurad, tablets, 200 mg + Zyloric®, allopurinol, tablet, 300 mg (comparator 1 + comparator 2).
  Interventions: Drug: lesinurad/allopurinol 200/300 FDC tablets; Drug: lesinurad 200 mg; Drug: allopurinol 300 mg
- Sequence BAAB (Experimental): Treatment A: Lesinurad/Allopurinol FDC Tablets - 200/300 mg (test product); Treatment B: lesinurad, tablets, 200 mg + Zyloric®, allopurinol, tablet, 300 mg (comparator 1 + comparator 2).
  Interventions: Drug: lesinurad/allopurinol 200/300 FDC tablets; Drug: lesinurad 200 mg; Drug: allopurinol 300 mg

INTERVENTIONS:
Drug: lesinurad/allopurinol 200/300 FDC tablets — Test Drug
Drug: lesinurad 200 mg — Comparator 1
Drug: allopurinol 300 mg — Comparator 2

SUMMARY:
To assess the bioequivalence between lesinurad/allopurinol 200/300 FDC tablets and coadministered lesinurad and allopurinol tablets in the fasted state based on the pharmacokinetic (PK) evaluation of lesinurad and allopurinol in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index ranging between 18.5 kg/m2 and 30 kg/m2.
* Screening serum urate level is ≤ 7.0 mg/dL.

Exclusion Criteria:

* Asian subject who has a positive test for the HLA-B*5801 allele.
* History or current diagnosis of kidney stones.
* Estimated creatinine clearance, as determined at Screening, of ≤ 80 mL/min calculated by the Cockcroft-Gault formula using ideal body weight.
* Undergone major surgery within 3 months prior to Screening.
* Donated blood within 4 weeks prior to Day 1 or experienced an event (other than blood donation) of significant blood loss (> 450 mL) within 12 weeks prior to Day 1 or has given a plasma donation within 4 weeks prior to Day 1.
* Inadequate venous access or unsuitable veins for repeated venipuncture.
* Received any strong or moderate enzyme-inducing drug or product within 2 months prior to Screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2017-10-04 (Actual); Study Completion 2017-10-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) endpoints in terms of maximum observed concentration (Cmax) for lesinurad/allopurinol 200/300 FDC tablets relative to lesinurad and allopurinol monocomponent tablets | Days 1, 8, 15 and 22
  Cmax is the maximum observed concentration of a drug after administration
PK endpoints in terms of area under the plasma concentration time curve from zero to the last quantifiable sampling timepoint (AUC last) for lesinurad/allopurinol 200/300 FDC tablets relative to lesinurad and allopurinol monocomponent tablets | Days 1, 8, 15 and 22
  AUC last is the area under the plasma concentration time curve from zero to the last quantifiable sampling timepoint
PK endpoints in terms of area under the plasma concentration time curve from and from zero to infinity (AUC 0-∞) for lesinurad/allopurinol 200/300 FDC tablets relative to lesinurad and allopurinol monocomponent tablets | Days 1, 8, 15 and 22
  AUC 0-∞ is a meausre of total concentration from time zero to infinity
PK endpoints in terms of time of occurrence of maximum observed concentration (tmax) for lesinurad/allopurinol 200/300 FDC tablets relative to lesinurad and allopurinol monocomponent tablets | Days 1, 8, 15 and 22
  Tmax is the time of occurrence of cmax
PK endpoints in terms of apparent terminal half-life (t1/2) for lesinurad/allopurinol 200/300 FDC tablets relative to lesinurad and allopurinol monocomponent tablets | Days 1, 8, 15 and 22
  t1/2 is a measure of apparent terminal half-life

SECONDARY OUTCOMES:
Incidence of Adverse Events in terms of changes in laboratory parameters | 26 days
Incidence of Adverse Events in terms of electrocardiogram parameters | 26 days
Incidence of Adverse Events in terms of vital signs | 26 days
Incidence of Adverse Events in terms of physical examination findings | 26 days

CONTACTS AND LOCATIONS:
Overall Officials: N. Bhakta, Study Director — Ardea Biosciences, Inc.
Locations (1):
- CAEP - Centro Avançado de Estudos e Pesquisas Ltda., Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No